CLINICAL TRIAL: NCT03169686
Title: The Efficacy of WeChat Based Interventions ('WeChat WeQuit' Program) for Smoking Cessation in China: a Randomized Trial
Brief Title: 'WeChat WeQuit' Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Attending Psychiatrist, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017S015
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Cigarette Smoking; Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive the 'WeChat WeQuit' program from the WeChat subscription account. The period for intervention was 14 weeks, including 2-week quiting preparation intervention and 12-week postquit intervention. The number of messages/pictures/audios received by participants will gradually decrease (will be intensively sent to them during 2-week prequit and 4-week postquit, and less intensively during 5-week to 12-week postquit), and follow-up questionnaires were sent only once a month in 14-28 weeks (week 16, 20, and 26 after the quit date). A WeChat group was created for answering questions from participants, and sharing the latest resources related to quitting smoking, and promoting communication between participants.
  Interventions: Behavioral: Cognitive and Behavioral Intervention
- Control Group (No Intervention): Control group participants will not receive any smoking cessation messages by professional team. They will receive messages of thanking them for being in the study and reminding them of the time until their free month at the end of follow up. In order to measure the main two outcomes (self-reported continuous smoking abstinence and point prevalence of abstinence), continuous smoking abstinence, point prevalence of abstinence, how many cigarettes per day during the last week if they are still smoking will be checked at week 1, 4, 8, 12, 16, 20 and 26 points.

INTERVENTIONS:
Behavioral: Cognitive and Behavioral Intervention — Participants who allocate to the intervention group will receive regular smoking cessation related information by professional team.
  Arms: Intervention Group

SUMMARY:
This proposed project is to assess whether WeChat-based smoking cessation interventions ('WeChat WeQuit' program) will be effective at helping people in China who smoke, to quit.

ELIGIBILITY:
Inclusion Criteria:

1. Daily Chinese cigarette smokers.
2. 18 years of age and older living.
3. Being able to read and write in Chinese.
4. Owning a smartphone and knowing how to use WeChat.
5. Willing to make an attempt to quit smoking in the next month.
6. Willing to provide informed consent to participate in the study.

Exclusion Criteria:

1. Nonsmokers.
2. Smokers without attempt to quit.
3. Below 18 years old.
4. Unable to use smartphone and WeChat.
5. Unable to read and write in Chinese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Biochemically Validated Continuously Abstinence | 26 weeks
  The primary outcome will be biochemical validation of self-reported 26-week continuous smoking abstinence

SECONDARY OUTCOMES:
Self-reported 7-day Point Abstinence | 26 weeks
  Self-reported 7-day point-prevalence abstinence at week 1, 4, 8, 12, 16, 20 and 26 after quit date.
Self-reported Continuous Abstinence | 26 weeks
  Self-reported continuous smoking abstinence rate at weeks 4, 8, 12, 16, 20, and 26 after the quit date.

OTHER OUTCOMES:
Smoking Reduction and Participation | 26 weeks
  Reductions in number of cigarettes smoked per day and rates of participation in and completion of smoking-cessation programs.

CONTACTS AND LOCATIONS:
Locations (1):
- Yanhui Liao, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (without personal information) will be included in submission and will be available to other researchers.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Tang J, Yang J, Liu Y, Liu X, Li L, Sun Y, Jin J, Fang Y, Zhou Z, Wang Y, Liu Y, Chen W, McNeill A, Kelly BC, Cohen JE, Liao Y. Efficacy of WeChat-based online smoking cessation intervention ('WeChat WeQuit') in China: a randomised controlled trial. EClinicalMedicine. 2023 May 18;60:102009. doi: 10.1016/j.eclinm.2023.102009. eCollection 2023 Jun. PMID 37251625